CLINICAL TRIAL: NCT06536868
Title: Tislelizumab Plus Chemotherapy and Concurrent Thoracic Radiotherapy as First-line Therapy for Extensive-stage Small-Cell Lung Cancer (ES-SCLC): an Multicenter, Single Arm Prospective Trial
Brief Title: Tislelizumab Combined With Chemotherapy and Thoracic Radiotherapy in ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Gang Jin, Dr., Second Hospital of Shanxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2024] YX No. 274
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tislelizumab; Etoposide; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICI+EC/EP+TRT (Experimental): Drug: Tislelizumab Drug: Carboplatin Drug: Etoposide Radiation: Radiation therapy Drug: Cisplatin
  Interventions: Drug: Tislelizumab; Drug: Etoposide; Drug: Carboplatin or Cisplatin; Radiation: Thoracic radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab infusion will be administered for 2 years (200mg, day1, Q3W).
Drug: Etoposide — Etoposide intravenous infusion will be administered during the induction phase (100mg/㎡, day1-3 Q3W for 4 cycles).
Drug: Carboplatin or Cisplatin — Carboplatin or Cisplatin intravenous infusion will be administered during the induction phase (Carboplatin AUC5, Q3W for 4 cycles; Cisplatin 75mg/㎡, Q3W for 4 cycles).
Radiation: Thoracic radiotherapy — IMRT 30-45Gy/10-15f

SUMMARY:
This study is a single arm, open, multicenter phase II study. The main purpose of this study was to evaluate preliminary efficacy and safety of Tislelizumab combined with thoracic radiotherapy as first line therapy for Extensive stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 80 years old (inclusive of 18th and 80th birthdays), male or female, at the time of signing the informed consent form;
* Confirmed small cell lung cancer of extensive stage by histology or cytology;
* At least one measurable lesion by imaging studies (according to RECIST 1.1) with a long diameter of ≥10 mm as examined by spiral CT or MRI;
* Within 3 days prior to treatment, an ECOG score of 0 to 1;
* No prior antitumor treatment for extensive stage disease (if the patient has previously received chemotherapy and/or radiotherapy in the limited stage of SCLC, the treatment intent must have been curative, and there must be at least a 6-month treatment-free interval between the end of chemotherapy, radiotherapy, or chemoradiotherapy and the diagnosis of extensive stage SCLC);
* Expected life span of ≥3 months;
* Good function of vital organs;
* The subject voluntarily joins this study, signs the informed consent form, has good compliance, and cooperates with follow-up.

Exclusion Criteria:

* Concurrent severe respiratory diseases: such as pulmonary fibrosis;
* Presence of psychiatric disorders, hematologic diseases, autoimmune diseases, and severe primary diseases of the heart, brain, liver, or kidneys;
* Uncontrolled active infections;
* Known or suspected allergies to the study medication and its excipients;
* Female patients who are pregnant or breastfeeding, or women of childbearing potential with a positive baseline pregnancy test;
* Prior use of antitumor treatment targeting the PD-(L)1 pathway.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 2 years
  From the date of enrollment to the date of disease progression

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR as assessed by the Investigator according to RECIST v1.1
Disease Control Rate (DCR) | Up to 2 years
  DCR as assessed by the Investigator according to RECIST v1.1
Overall Survival （OS） | Up to 2 years
  From the date of enrollment until death by any cause or last follow-up
Adverse events | Up to 2 years
  Treatment-related adverse events according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Dr., Principal Investigator — Second Hospital of Shanxi Medical University
Locations (6):
- China (6):
  - Jincheng General Hospital, Jincheng, Shanxi
  - Jinzhong third people's hospital, Jinzhong, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Hospital of Traditional Chinese Medicine, Taiyuan, Shanxi
  - TISCO General Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No